CLINICAL TRIAL: NCT01016834
Title: A Multicenter, Open-label Evaluation of Treatment Satisfaction, Tolerability, Safety and Preference for Sumavel DosePro for Treatment of Migraine in Subjects Currently Treated With Triptans
Brief Title: Evaluation of Treatment Satisfaction and Preference for Sumavel DosePro in the Treatment of Migraine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zogenix, Inc. (Industry)
Collaborators: Synteract, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZX001-0901
Record Dates: First submitted 2009-11-18; First posted 2009-11-20 (Estimated); Results first posted 2011-12-29 (Estimated); Last update posted 2011-12-29 (Estimated); Status verified 2011-11

CONDITIONS: Migraine
Keywords: migraine; treatment satisfaction
MeSH Terms: conditions — Migraine Disorders | interventions — Sumatriptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sumavel(R) DosePro(R) (Other): Single arm study (Sumavel DosePro)
  Interventions: Device: Sumavel DosePro; Drug: Sumatriptan

INTERVENTIONS:
Device: Sumavel DosePro — Needle free delivery system containing 0.5 mL of solution of 6 mg sumatriptan, subcutaneous administration
Drug: Sumatriptan — subcutaneous injection, 6 mg, per migraine attack, no more than two administrations within a 24 hr period
  Other Names: Sumavel DosePro (Sumatriptan injection)

SUMMARY:
The purpose of the study is to evaluate the treatment satisfaction of subjects using Sumavel DosePro to treat their moderate to severe migraines.

DETAILED DESCRIPTION:
Single arm, open-label, multicenter study to evaluate the treatment satisfaction, treatment confidence, and subject preference for Sumavel DosePro in adult subjects diagnosed with migraines and currently treated with triptans. Subjects will treat up to 4 migraines over a 60 day period and complete migraine diaries and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* History of 2 to 6 migraine headaches per month
* Migraines should have been present for at least 1 year with age at onset of migraine less than 50 years
* History of 24 hours of freedom between migraine attacks
* Current users of triptan medications
* Able to distinguish interval or other non-migrainous headaches from typical migraine
* General good health

Exclusion Criteria:

* History or symptoms, or signs of ischemic cardiac, cerebrovascular, or peripheral vascular syndromes
* Significant underlying cardiovascular diseases including uncontrolled hypertension
* Hemiplegic or basilar migraine
* History or diagnosis of severe hepatic or renal impairment
* History of epilepsy or seizure or other serious neurologic condition
* History of allergy, anaphylaxis, or hypersensitivity to sumatriptan or any of its components or similar drugs including sulphonamides
* History of scleroderma (systemic sclerosis)
* Pregnant or breastfeeding
* Use of contraindicated prescription medications, monoamine oxidase inhibitors (MAO-A), selective serotonin reuptake inhibitors, or lithium agents

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2009-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger K Cady, MD, Study Chair — Clinvest
Locations (21):
- United States (21):
  - University of Alabama Hospital, Dept. of Neurology, Birmingham, Alabama
  - Arizona Research Center, Phoenix, Arizona
  - C. Phillip O'Carroll, MD, Inc, Newport Beach, California
  - California Medical Clinic for Headache, Santa Monica, California
  - Alpine Clinical Research, Boulder, Colorado
  - University Clinical Research Inc., Pembroke Pines, Florida
  - Comprehensive Neuroscience Inc, St. Petersburg, Florida
  - Comprehensive Neurosciences Inc, Atlanta, Georgia
  - Neurology Specialists of Decatur, Decatur, Georgia
  - Diamond Headache Clinic, Chicago, Illinois
  - Michigan Head, Pain, & Neurological Institute, Ann Arbor, Michigan
  - Clinvest/A Division of Banyan Group, Inc, Springfield, Missouri
  - Mercy Health Research, St Louis, Missouri
  - Meridian Clinical Research, Omaha, Nebraska
  - Regional Clinical Research Inc, Endwell, New York
  - Headache Wellness Center, Greensboro, North Carolina
  - Cleveland Clinic: Neurological Center for Pain, Cleveland, Ohio
  - Jefferson Headache Center, Philadelphia, Pennsylvania
  - Neurological Medicine, Clarksville, Tennessee
  - Nashville Neuroscience Group, Nashville, Tennessee
  - Swedish Pain and Headache Center, Seattle, Washington

REFERENCES:
- [Derived] Rothrock JF, Cady RK, Aurora SK, Brandes JL, Myers JA, Fox AW, Farr SJ. Needle-free subcutaneous sumatriptan for triptan users requiring a change in migraine therapy: efficacy and impact on patient-rated functionality, satisfaction, and confidence. Curr Med Res Opin. 2011 Nov;27(11):2185-91. doi: 10.1185/03007995.2011.619177. Epub 2011 Sep 26. PMID 21942531
- [Derived] Cady RK, Aurora SK, Brandes JL, Rothrock JF, Myers JA, Fox AW, Farr SJ. Satisfaction with and confidence in needle-free subcutaneous sumatriptan in patients currently treated with triptans. Headache. 2011 Sep;51(8):1202-11. doi: 10.1111/j.1526-4610.2011.01972.x. Epub 2011 Aug 3. PMID 21812775

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period occured from November, 2009 to February, 2010 at 22 US medical clinics
Groups:
- Sumavel DosePro: The primary study endpoint was overall subject satisfaction with Sumavel DosePro, based on a comparison of the subject's self-reported answer to the single overall satisfaction question completed at the beginning of the study based on his or her pre-study triptan treatment versus at the end of their treatment period.
Period: Overall Study
Arm/Group | Sumavel DosePro
Started | 242
Completed | 220
Not Completed | 22

BASELINE CHARACTERISTICS:
Arm/Group | Sumavel DosePro
Number analyzed (Participants) | 242
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 242
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 196
  Male | 46
Region of Enrollment [Number; unit: participants]
  United States | 242

OUTCOME MEASURES:

1. Primary Outcome: Overall Satisfaction
Description: Change from baseline in overall subject satisfaction with migraine treatments. Patient Perception of Migraine Questionnaire-Revised, question 3c "Overall satisfaction" was the measure. Baseline measured subjects satisfaction with past migraine treatments. End of study measured subject's satisfaction with migraine treatment by Sumavel DosePro. PPMQ-R scale (1-7 scale; 1=very satisfied)is transformed to a 0-100 scale (100=very satisfied)
Time Frame: After 4 migraines or 60 days
Population: The Per-protocol (PP) population included all subjects who treated at least one (and up to four) migraine episode(s) with Sumavel DosePro and complied with all other study procedures.
Measure: Mean (Standard Deviation); unit: Scale of 0-100; 100= very satisfied
Arm/Group | Sumavel DosePro
Number analyzed (Participants) | 211
Scale of 0-100; 100= very satisfied | 73.7 (29.08)
Statistical Analysis 1: Comparison: Sumavel DosePro; For the primary analyses and other PPMQ-R variables, the mean of the differences between each subject's rating of overall treatment satisfaction at the end of study based on the subject's experience using Sumavel DosePro and the rating at baseline based on the subject's pre-study triptan treatment were compared using a two-sided paired t-test at the 5% level of significance; Test type: Superiority or Other; p = 0.0007, t-test, 2 sided

2. Secondary Outcome: Treatment Preference
Description: Number of subjects preferring Sumavel DosePro compared to their pre-study migraine treatment (Prefer Sumavel DosePro vs. No Preference or Prefer Other Treatment).
Time Frame: After 4 migraines or 60 days
Measure: Number; unit: participants
Arm/Group | Sumavel DosePro
Number analyzed (Participants) | 211
participants | 74 [29.6 to 40.8]

3. Secondary Outcome: Treatment Confidence
Description: Number of subjects who indicated they were confident or very confident in treating repeated migraine attacks with Sumavel DosePro at end of treatment.
Time Frame: After 4 migraines or 60 days
Measure: Number; unit: participants
Arm/Group | Sumavel DosePro
Number analyzed (Participants) | 211
participants | 136

ADVERSE EVENTS:
Time Frame: 60 days
Description: Subjects were asked to report SAEs from first dose of Sumavel DosePro up to 3-5 days post 4th migraine attack or 60 days, which ever occurred earliest.
Arm/Group | Sumavel DosePro
Serious Adverse Events (participants affected / at risk) | 0/242
Other Adverse Events (participants affected / at risk) | 136/242
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sumavel DosePro (N=242)
Administrative site conditions (General disorders) | 99 — Inclusive of all single reports of injection site hemorrhage,hematoma, pain, swelling, and erythema
Dizzyness (Nervous system disorders) | 17
Paresthesia (Nervous system disorders) | 14
Somnolence (Nervous system disorders) | 13
Nausea (Gastrointestinal disorders) | 18
Dry mouth (Gastrointestinal disorders) | 12
Muscle tightness (Musculoskeletal and connective tissue disorders) | 14
Flushing (Vascular disorders) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days